CLINICAL TRIAL: NCT02982343
Title: BALTiC Study: A Feasibility Analysis of Home Based BALance Training in People With Charcot-Marie-Tooth Disease
Acronym: BALTiC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Collaborators: Charcot Marie Tooth United Kingdom (Unknown); Kingston University (Other)
Responsible Party: Principal Investigator, Gita Ramdharry, Principle Investigator, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/LO/0720
Record Dates: First submitted 2016-11-28; First posted 2016-12-05 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Charcot-Marie-Tooth Disease, Type IA
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Falls management plus exercise training (Experimental): Falls management and education session. Home proximal lower limb strength training and multi-sensory balance training.
  Interventions: Behavioral: Falls management plus exercise training
- Falls management only (Active Comparator): Falls management and education session only.
  Interventions: Behavioral: Falls management only

INTERVENTIONS:
Behavioral: Falls management plus exercise training — Participants will undergo a session of falls management and education followed by 12 weeks of strength and balance training. Strength training will be performed 4 times per week. Resistance training of the proximal muscles will be prescribed progressing to loads of 60% of 1 repetition maximum, 8-12 repetitions. Weaker muscles will be trained using 2 sets of 8-12 repetitions against gravity. They will also give a selection of exercises targeting balance to challenge stability and sensory feedback using equipment such as foam cushions, though will be individual based on participants' limitations and abilities. Participants will be asked to perform balance exercises daily.
  Arms: Falls management plus exercise training
Behavioral: Falls management only — Participants will undergo a session of falls management and education.
  Arms: Falls management only

SUMMARY:
Charcot Marie Tooth (CMT) is the most common inherited neuropathy. It affects the nerves of the hands and feet first, slowly progressing towards the centre of the body. It causes varying degrees of weakness and reduced feeling, usually affecting the feet and ankles first. High incidence of falls and knock on effects in quality of life are common. This is a lifelong condition which, though not life limiting, does not have a cure. Research into the effect of balance rehabilitation in people with CMT has been limited to traditional exercises, which do not address the complex nature of balance impairments in this condition. Multi-sensory rehabilitation has proved beneficial in improving balance in people with sensory neuropathy. Research shows that strengthening trunk muscles can improve balance in older people. Trunk and muscles close to it are largely unaffected in people with CMT, therefore these muscles could be strengthened in these patients. This study proposes to assess the feasibility of multi-sensory balance training, strength training with a focus on the trunk and muscles close to the trunk, and falls management education. This comprehensive approach is reflective of a clinical physiotherapy programme. Though a life-long condition, many people with CMT lead full lives. A home based programme is proposed to so that patients can fit it into their lives without having to travel for treatment. Therapists will use self-management principles within treatment. Measurements will be taken prior to and following treatment including physical measures, questionnaires and interviews. The physiotherapy interventions will be taught home and data collection will be at the National Hospital for Neurology and Neurosurgery, University College London Hospitals (UCLH).

DETAILED DESCRIPTION:
A recent, unpublished focus group study of people with CMT found that they reported more falls than healthy people. They reported problems walking on uneven surfaces, difficulty getting off the floor and a necessity to consciously think about every step to avoid falling while walking (GM Ramdharry et al., 2015). A retrospective survey of people with CMT found that 89% of the 94 respondents reported falls to the ground. Half of them reported falling at least once a month with 5% falling every day (Ramdharry et al., 2011). We have just completed an exploratory study of factors predicting falls risk. Preliminary analysis of prospective falls data for 32 people over 6 months showed that they fell a median of 4 times (range 0 - 54 falls) and functional balance performance may be predictive (Ramdharry et al., 2015). A study of people with CMT1a found that sensory impairment increased visual dependence for a static balance task (van der Linden et al., 2010). There has only been one small study of balance training in people with CMT, comparing a novel rehabilitation device with more traditional exercises (Matjacić and Zupan, 2006). Both interventions showed improvement in functional balance scores. Studies of proximal strength training in CMT have shown improvements in walking parameters (Chetlin et al., 2004; Lindeman et al., 1995), but the effect on balance has not been explored. Because of the mixed sensori-motor presentation of people with CMT, a combined approach of multi-sensory balance training and proximal strengthening will be delivered. A home-based model has been proposed as CMT is a life-long condition that needs to be managed by the individual outside of the medical or therapy environment.

STUDY DESIGN & JUSTIFICATION A single blinded randomised controlled design has been chosen in this feasibility study. The intention is to see if there is an effect of the intervention to later be explored in a larger randomized controlled trial. A blinded assessor will measure balance performance prior to randomisation and following the 12 weeks of either intervention or control. They will also undertake qualitative interviews prior to randomization and following final measurement session. Interviews will inform the intervention and its acceptability. All participants will receive a falls assessment and falls education. Following randomisation, participants will either receive the 12-week intervention or control period. The intervention will include a holistic programme of physiotherapy including strength training of muscle groups unaffected by the condition and multi-sensory exercises to target balance. The program will be delivered by a physiotherapist trained in delivering treatment under the principles of self-management. Exercises will be carried out by the patients in their own homes and monitored by the research physiotherapist, progressing as appropriate. Those randomized to the control arm will receive monitoring telephone calls throughout this 12-week period.

RECRUITMENT Patients will be recruited from outpatient neurology clinics at Queen Square which specialise in the diagnosis and management of CMT. Patients who fit the inclusion criteria will be approached and the trial will be described to them. Written information will be provided and arrangement made for a way to make contact once they have decided about whether they wish to proceed with screening. All patients who agree to proceed will go through a screening which will take place over the telephone. Those who pass screening will be provided with falls diary postcards or arrangement for falls diary emails, which they will be asked to monitor and report for one month. A sample will be invited for a qualitative interview. Arrangement will be made for them to attend a baseline measurement session, falls assessment, and falls education following the month-long falls monitoring.

Measures will include:

Patient reported questionnaires of balance confidence, mood, walking ability and physical functioning 10m walk test / 6 minute walk test Berg Balance Scale Bruininks Oseretsky Test (BOT) BESTest Functional balance tests using force plate and movement analysis equipment Strength testing of the lower limbs and hands Charcot Marie Tooth Examination Score (CMTES) A block randomisation will occur following the baseline measurement and falls education session with allocation either being to a control arm or an intervention arm. This will be done by the PI or research physiotherapist who will remain un-blinded. Contact with the blinded assessor will cease until the final measurement session 12 weeks later.

INTERVENTION:

If randomised to the control arm of the study, participants will be advised that the research physiotherapist will contact them monthly to monitor any falls or issues. For those randomised to the intervention arm, a home visit will be arranged with the research physiotherapist as soon as possible. During this session, the research physiotherapist will provide the participant with exercises to strengthen the muscles of the trunk and proximal muscles using body weight and graded ankle weights. Strength training will be performed 4 times per week. They will also give a selection of exercises targeting balance to challenge stability and sensory feedback. Participants will be asked to perform balance exercises daily. A risk assessment will be undertaken with guidance on how to ensure safety when doing the exercises. An exercise diary will be provided for the participants to monitor exercise frequency.

Arrangements will be made for weekly telephone calls with the research physiotherapist to monitor progress and a provisional date set for the first monthly home monitoring visit. Participants in the intervention arm will be contacted weekly for 12 weeks on the study. The research physiotherapist will visit them at home to monitor and progress exercises once a month during this time.

QUALITATIVE RESEARCH At the consent meeting all patients will be invited to take part in interviews conducted after the consent meeting and following completion of the final measurements. They will be made aware that participation in the interviews is supplementary to the main study and they are free to decline. Purposive sampling will be used to ensure a sample of maximum diversity of age, gender, and symptom severity. Potential qualitative interview participants will be given written details of the qualitative study and asked to give their consent to be interviewed if they are willing to take part. The interview will be audio recorded and consist of a dialogue between the interviewer (the researcher) and the participant. A topic guide will be used during the interviews, but the participant will be invited to raise issues of importance to them. Data analysis will be iterative, in that it will be continually analysed throughout the data collection process and used to inform following interviews.

PROCEDURES TO DEAL WITH RESEARCHER EFFECTS AND BIAS Assessments will be carried out by a blinded assessor to standardise treatment during tests. Falls assessment and falls education will be provided at the baseline measurement session by the blinded assessor, prior to participant randomisation. In this way participants will be given the same treatment. The blinded assessor will perform final measurements. The participant will be reminded prior to the start the final session to not mention what they may or may not have been doing in the 12 weeks prior to maintain blinding throughout the session

ELIGIBILITY:
Inclusion Criteria:

1. Genetically confirmed diagnosis of CMT1a
2. History of falls
3. Mixed sensory and motor presentation
4. Over 18 years
5. Able to stand unsupported for five minutes
6. Able to walk for 50m with or without a walking stick or orthotic devices

Exclusion Criteria:

1. Presence of other significant neurological disorders (such as multiple sclerosis, cerebrovascular diseases, epilepsy, movement disorders), or major comorbidities (e.g. vestibular dysfunction, use of medication which may affect balance, cognitive impairment, presence of medical conditions in which exercise training may be detrimental).
2. Presence of peripheral neuropathy caused by a condition other then CMT.
3. Limb surgery during the six months prior to screening (or planned before final assessment).
4. Participation in any other concurrent intervention trial, or less than six months after cessation of an intervention trial.
5. Women of child-bearing age if they are pregnant, planning a pregnancy during their time in the study or in the 12 weeks following giving birth. This is due to the effects of pregnancy on balance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Balance performance | 12 weeks
  Balance performance will be measured using laboratory measures of postural stability during static and dynamic tasks. Centre of pressure excursion and velocity will be the main variables

SECONDARY OUTCOMES:
Recruitment rate | 1 year
  For this feasibility study, recruitment rate data will be gathered
Falls monitoring | 20 weeks
  Falls monitoring will be done one month before, during the 12 week invention/control period and one month afterwards using postcards or a web based app, depending on participant preference.
Bruininks Oseretsky Test (BOT) | 12 weeks
  Clinician rated measure of functional balance performance.
Berg Balance test | 12 weeks
  Clinician rated measure of functional balance performance.
BESTest | 12 weeks
  Clinician rated measure of functional balance performance.
10 minute timed walk | 12 weeks
  Walking speed test
Quantitative lower limb muscle strength testing | 12 weeks
  Hand-held myometry protocol performed by rater for the major lower limb muscle groups.
CMTES: Charcot Marie Tooth Examination Score | 12 weeks
  Clinician rated disease severity scale
Falls Self Efficacy Scale | 12 weeks
  Patient reported outcome measure of balance confidence. Questionnaire.
Walk-12 | 12 weeks
  Patient reported outcome measure of walking function. Questionnaire.
IPAQ: International Physical Activity Questionnaire | 12 weeks
  Patient reported outcome measure of physical activity. Questionnaire.
SF36: Short Form 36 | 12 weeks
  Patient reported outcome measure of health related quality of life. Questionnaire.
Hospital Anxiety and Depression Score | 12 weeks
  Patient reported outcome measure of depression and anxiety symptoms. Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gita M Ramdharry, PhD, Principal Investigator — University College London Hosptials NHS Trust
Locations (1):
- National Hospital for Neurology and Neurosurgery, UCLH, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramdharry, G., M. Dudziec, D. Tropman, E. Dewar, A. Wallace, M. Laura, R. Grant, and M. Reilly. 2015. 'Exploring the Causes of Falls and Balance Impairments in People with Charcot-Marie Tooth Disease'. Physiotherapy 101 (May): e1255. doi:10.1016/j.physio.2015.03.1159.
- [Background] Ramdharry GM, Pollard A, Anderson C, Laura M, Murphy SM, Dudziec M, Dewar EL, Hutton E, Grant R, Reilly MM. A pilot study of proximal strength training in Charcot-Marie-Tooth disease. J Peripher Nerv Syst. 2014 Dec;19(4):328-32. doi: 10.1111/jns.12100. PMID 25582960
- [Background] van der Linden MH, van der Linden SC, Hendricks HT, van Engelen BG, Geurts AC. Postural instability in Charcot-Marie-Tooth type 1A patients is strongly associated with reduced somatosensation. Gait Posture. 2010 Apr;31(4):483-8. doi: 10.1016/j.gaitpost.2010.02.005. Epub 2010 Mar 11. PMID 20226674
- [Background] Matjacic Z, Zupan A. Effects of dynamic balance training during standing and stepping in patients with hereditary sensory motor neuropathy. Disabil Rehabil. 2006 Dec 15;28(23):1455-9. doi: 10.1080/09638280600646169. PMID 17166808
- [Background] Chetlin RD, Gutmann L, Tarnopolsky M, Ullrich IH, Yeater RA. Resistance training effectiveness in patients with Charcot-Marie-Tooth disease: recommendations for exercise prescription. Arch Phys Med Rehabil. 2004 Aug;85(8):1217-23. doi: 10.1016/j.apmr.2003.12.025. PMID 15295743
- [Background] Lindeman E, Leffers P, Spaans F, Drukker J, Reulen J, Kerckhoffs M, Koke A. Strength training in patients with myotonic dystrophy and hereditary motor and sensory neuropathy: a randomized clinical trial. Arch Phys Med Rehabil. 1995 Jul;76(7):612-20. doi: 10.1016/s0003-9993(95)80629-6. PMID 7605179